CLINICAL TRIAL: NCT03730805
Title: The Adaptation and Evaluation of the WHO's ASSIST-linked Brief Intervention to Khat-Using Ethiopian University Students
Acronym: KhatAssist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Jimma University (Other)
Responsible Party: Principal Investigator, Michael Odenwald, Managing Director, Outpatient Clinic for Psychotherapy, University of Konstanz
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: KHAT ASSIST 2018
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Khat Abuse
Keywords: Catha Edulis; Khat; Qat; Khat Use Disorder; Screening and Brief Intervention; ASSIST
MeSH Terms: conditions — Helping Behavior | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Intervention + open mindset (Experimental): ASSIST-linked Brief Intervention plus prior induction of deliberative mindset
  Interventions: Behavioral: ASSIST-linked Brief Intervention; Behavioral: Induction of Deliberative Mindset
- Intervention + closed mindset (Experimental): ASSIST-linked Brief Intervention plus prior induction of closed mindset
  Interventions: Behavioral: ASSIST-linked Brief Intervention; Behavioral: Induction of Implemental Mindset
- Intervention alone (Experimental): ASSIST-linked Brief Intervention without prior induction of any mindset
  Interventions: Behavioral: ASSIST-linked Brief Intervention
- Control + open mindset (Experimental): In stead of intervention, a neuropsychological assessment (Raven's Standard Progressive Matrices; SPM; Raven, 1940) with prior induction of an open mindset is conduced.
  Interventions: Behavioral: Induction of Deliberative Mindset
- Control + closed mindset (Experimental): In stead of intervention, a neuropsychological assessment (Raven's Standard Progressive Matrices; SPM; Raven, 1940) with prior induction of a closed mindset is conduced.
  Interventions: Behavioral: Induction of Implemental Mindset
- Control alone (No Intervention): In stead of intervention, a neuropsychological assessment (Raven's Standard Progressive Matrices; SPM; Raven, 1940) without prior induction of any mindset is conduced.

INTERVENTIONS:
Behavioral: ASSIST-linked Brief Intervention — The intervention follows the WHO's ASSIST-linked Brief Intervention (Humenik et al., 2012; Humeniuk et al., 2010), a manualized one-session intervention that can be categorised as belonging to the Screening and Brief Intervention approach. It follows the FRAMES model (Bien et al., 1993) and contains techniques from Motivational Interviewing (Miller & Rollnick, 1991).
  Other Names: Screening and Brief Intervention
  Arms: Intervention + closed mindset; Intervention + open mindset; Intervention alone
Behavioral: Induction of Deliberative Mindset — Based on the Mindset Theory of Action Phases (Gollwitzer & Keller, 2016), a brief writing task (writing down pros and cons for an unresolved personal problem of the participant's own choice) is used to induce a specific psychological state in which the individual is cognitively open to process new information.
  Other Names: Induction of Open Mindset
  Arms: Control + open mindset; Intervention + open mindset
Behavioral: Induction of Implemental Mindset — Based on the Mindset Theory of Action Phases (Gollwitzer & Keller, 2016), a brief writing task (writing down steps necessary to implement a personal decision of the participant's choice that has not yet been put into practice) is used to induce a specific psychological state in which the individual is cognitively not open to process new information.
  Other Names: Induction of Closed Mindset
  Arms: Control + closed mindset; Intervention + closed mindset

SUMMARY:
The leaves of the khat tree (catha edulis) are traditionally chewed in the countries around the Horn of Africa. They contain the amphetamine-like alkaloid cathinone and their use can produce a Substance Use Disorder. The researchers intent to validate an Amharic and an Oromo version of the WHO's ASSIST-linked Brief Intervention among khat-using Ethiopian university students. In an RCT, khat using students of Jimma University with initial motivation to stop or cut down khat use will be randomised to either an intervention or a control group. In the intervention group, the WHO's ASSIST-linked BI will be delivered in a single session by trained local counsellors. In the control group, participants will receive a neuropsychological assessment (Raven's Standard Progressive Matrices, SPM; Raven, 1972). Khat use, the neuropsychological variables and psychiatric symptoms will be assessed before the intervention and two weeks after it. Additionally, the researchers will measure the participants resistance during the session. The control group will receive the intervention after the post test. In order to study state variables that influence brief intervention effectivity, e.g. by increasing or reducing resistance, the researchers randomise subjects in each study arm to several short pre-interventions that are based on Gollwitzer's empirically well established Mindset Theory of Action Phases (for summary: Gollwitzer & Keller, 2016). This means, before delivering the ASSIST-linked BI (intervention group) or before the SPM assessment (controlgroup) a specific psychological state will be induced by a brief writing task that theoretically should affect the openness to the intervention: (1) implemental mindset, (2) deliberative mindset, (3) no mindset induction. The researchers expect that khat use will be reduced more in the intervention condition compared to the control condition and that induced states influence the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* second year student or higher year student at Jimma University
* khat use in the month prior to baseline
* participant's wish to reduce or stop khat use

Exclusion Criteria:

* severe substance use, except khat
* inability to read and write Amharic or Oromo languages
* ongoing acute episode of severe mental disorder
* current suicidal ideation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 307 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
khat use quantity (standard units) | Change from T1 (Baseline at study entry) to T2 (two weeks after ASSIST-linked BI (intervention group) or two weeks after baseline assessment (control group))
  The researchers assess the khat units consumed in the two weeks prior to the assessment with Sobell & Sobell's (1995) calender-based method, Timeline Follow Back.
days with khat use | Change from T1 (Baseline at study entry) to T2 (two weeks after ASSIST-linked BI (intervention group) or two weeks after baseline assessment (control group))
  The researchers assess the days with khat use in the two weeks prior to the assessment with Sobell & Sobell's (1995) calender-based method, Timeline Follow Back.

SECONDARY OUTCOMES:
Problem solving | Change from T1 (Baseline at study entry) to T2 (two weeks after ASSIST-linked BI (intervention group) or two weeks after baseline assessment (control group))
  The researchers use the Tower of Hanoi to assess the ability of the individual to solve a problem. Time to solve the problem in seconds sis recorded.
Working memory | Change from T1 (Baseline at study entry) to T2 (Two weeks after ASSIST-linked BI (intervention group) or two weeks after baseline assessment (control group))
  The researchers use the Corsi Block Tapping Task (Corsi, 1972) to assess the visio-spacial working memory performance of the respondent.
Symptoms of depression and anxiety | Change from T1 (Baseline at study entry) to T2 (two weeks after ASSIST-linked BI (intervention group) or two weeks after baseline assessment (control group))
  The researchers use the sum scale of the Self-Report Questionnaire 20 (SRQ-20; Harding et al., 1983) to measure symptoms of depression and anxiety.
Symptoms of khat-induced psychosis | Change from T1 (Baseline at study entry) to T2 (two weeks after ASSIST-linked BI (intervention group) or two weeks after baseline assessment (control group))
  The researchers use four items from the WHO's Composite International Clinical Interview (CIDI) to assess khat-induced psychotic symptoms according to the procedure published by Widmann et al. (2014).
Resistance during intervention session | Immediately after the intervention session (ASSIST-linked BI) or control session (SPM assessment)
  Counsellors rate the participants degree of cooperativeness and resistance with the method developed by Haller et al. (2018).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Odenwald, PhD, Principal Investigator — University of Konstanz
Locations (1):
- Jimma University, Jimma, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gollwitzer, P., & Keller, L. (2016). Mindset Theory. In V. Zeigler-Hill & T. K. Shackleford (Eds.), Encyclopedia of Personality and Individual Differences. New York: Springer.
- [Background] Corsi, P. M. (1972). Human memory and the medial temporal region of the brain. Dissertation Abstracts International, 34, 819B.
- [Background] Harding TW, Climent CE, Diop M, Giel R, Ibrahim HH, Murthy RS, Suleiman MA, Wig NN. The WHO collaborative study on strategies for extending mental health care, II: The development of new research methods. Am J Psychiatry. 1983 Nov;140(11):1474-80. doi: 10.1176/ajp.140.11.1474. PMID 6624995
- [Background] Humeniuk R, Ali R, Babor T, Souza-Formigoni ML, de Lacerda RB, Ling W, McRee B, Newcombe D, Pal H, Poznyak V, Simon S, Vendetti J. A randomized controlled trial of a brief intervention for illicit drugs linked to the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) in clients recruited from primary health-care settings in four countries. Addiction. 2012 May;107(5):957-66. doi: 10.1111/j.1360-0443.2011.03740.x. Epub 2012 Feb 28. PMID 22126102
- [Background] Humeniuk, R., Henry-Edwards, S., Ali, R., Poznyak, V., Monteiro, M., & World Health Organization. (2010). The ASSIST-linked Brief Intervention for Hazardous and Harmful Substance Use: Manual for Use in Primary Care. Geneva: World Health Organization.
- [Background] Miller, W. R., & Rollnick, S. (1991). Motivational interviewing : preparing people to change addictive behavior. New York: Guilford Press.
- [Background] Widmann M, Warsame AH, Mikulica J, von Beust J, Isse MM, Ndetei D, al'Absi M, Odenwald MG. Khat Use, PTSD and Psychotic Symptoms among Somali Refugees in Nairobi - A Pilot Study. Front Public Health. 2014 Jun 30;2:71. doi: 10.3389/fpubh.2014.00071. eCollection 2014. PMID 25072043
- [Background] Sobell, L. C., & Sobell, M. B. (1995). Alcohol Timeline Followback Users's Manual. Toronto: Addiction Research Foundation.
- [Background] Bien TH, Miller WR, Tonigan JS. Brief interventions for alcohol problems: a review. Addiction. 1993 Mar;88(3):315-35. doi: 10.1111/j.1360-0443.1993.tb00820.x. PMID 8461850
- [Background] Raven JC. Matrix Tests. Ment Health (Lond). 1940 Jan;1(1):10-18. No abstract available. PMID 28908970
- [Background] Haller, N., Keller, L., Treiber, J., Schrietter, F., & Odenwald, M. (2018). The effect of mindset inductions on motivational interventions to reduce alcohol use: a pilot studies among university students. Poster presentation at the German Addiction Conference, September 17 - 20, 2018, Hamburg, Germany.